CLINICAL TRIAL: NCT03515759
Title: The Efficacy of Fetal Arterial and Venous Doppler Indices in Predicting Perinatal Outcome Among Severely Hypertensive Pregnant Patients.
Brief Title: Fetal Doppler Indices in Predicting Perinatal Outcome Among Severely Hypertensive Pregnant Patients.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, assistant professor, Cairo University
Other Study IDs: 2062010
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-04

CONDITIONS: Pre-Eclampsia; IUGR
Keywords: PREECLAMPSIA; DOPPLER; IUGR; UMBILICAL ARTERY; MIDDLE CEREBRAL ARTERY
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hypertensive patients: 60 pregnant women with singleton living fetus between 34 -38 wks gestation known to have severe hypertension in the current pregnancy were included

SUMMARY:
60 pregnant women with singleton living fetus between 34 -38 wks gestation known to have severe hypertension in the current pregnancy were included.

All participants underwent Doppler ultrasonography to evaluate the Feto-Placental Circulation within 24 hours from Pregnancy Termination.

Flow Velocity Waveforms were obtained from: Umbilical Artery (UA), Middle Cerebral Artery (MCA), Ductus Venosus (DV), Umbilical Vein (UV).

From the flow velocity waveforms the following indices were measured:

UA & MCA: Pulsatility Index (PI) & Resistance Index (RI), DV: Peak Velocity Index For veins (PVIV), Peak Systolic Velocity (PSV) & a- wave.

UV Flow: Presence or Absence of Pulsatile Flow.

DETAILED DESCRIPTION:
60 pregnant women (aged from 18- 35 years) with singleton healthy living fetus between 34 -38 wks gestation known to have severe hypertension in the current pregnancy were included.

Chronic Hypertension was defined as a blood pressure value of 140/90 mm Hg or higher diagnosed before 20 weeks' gestation or preconception. Gestational Hypertension was defined as blood pressure value of 140/90 mm Hg or higher on 2 occasions at least 4 hours apart that occurred after 20 weeks' gestation in a patient with previously normal blood pressure. Preeclampsia was defined as blood pressure value of 140/90 mm Hg or higher on 2 occasions at least 4 hours apart and proteinuria (Proteinuria is defined as the excretion of 300mg or more of protein in a 24 hour urine collection or 1+ by The dipstick method) that occurred after 20 weeks' gestation in a patient with previously normal blood pressure. Chronic hypertension & gestational hypertension was considered to be severe if systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥110 mmHg, or both & persists for 15 minutes or more. Preeclampsia was considered to be severe in the following conditions: Blood pressure of 160/110 or more, Thrombocytopenia (platelet count less than 1000,000 / microliter), impaired liver function (elevated blood levels of liver transaminases to twice the normal concentration) , severe persistent right upper quadrant or epigastric pain unresponsive to medication and not accounted for by alternative diagnosis, or both, the new development of renal insufficiency (elevated serum creatinine > 1.1mg/dL or a doubling of serum creatinine in the absence of other renal disease) & new-onset cerebral or visual disturbances. Patients with other maternal medical disorders rather than hypertension or experienced rupture of membrane or antepartum hemorrhage (placenta previa or accidental hemorrhage) were excluded. Also, patients who received respiratory depressants medications within 2 hours from the delivery of the fetus (e. g., opioid analgesic) were excluded.

Informed consents were obtained from all participants after explanation of the study and its aims. All participants underwent the following: Full history taking including a detailed history of the hypertension state during the current pregnancy (onset, course, current medication, and whether the blood pressure is controlled or not). complete physical examination: general (including BMI & blood pressure measurement) and obstetric examinations. Routine obstetric ultrasound: to confirm gestational age & fetal viability & number, assess fetal weight (EFW) and growth percentile & amniotic fluid index (AFI) & to exclude fetal anomalies. Laboratory investigations (Complete blood count (CBC) - Urine analysis for albuminuria - Liver enzymes & kidney function). In addition to Doppler ultrasonography assessment using GE Voluson Pro-V and GE Voluson E10 with 3.5-5 MHz abdominal transducer). The color flow imaging (to identify the vessels) & pulsed wave velocimetry was used to obtain flow velocity waveforms within 24 hours of pregnancy termination from: Umbilical artery (UA): from a free-floating loop in the mid portion of the cord, Middle cerebral artery (MCA): obtained from a transverse image of the fetal head at the level of sphenoid bones (color flow im¬aging was used to display the circle of Willis), Ductus venosus (DV) was sampled soon after its origin from the umbilical vein & finally Umbilical vein flow (UV) assessment. In all Doppler studies, while the woman is lying in a semi-recumbent position, the angle of insonation of the vessels is < 45 degrees & the high-pass filter is set at 100 Hz. Care is taken not to exert undue pressure on the fetal head because this alters the flow velocity waveforms from the MCA. Furthermore, examination of the fetal vessels was performed in the absence of fetal body and respiratory movements, with a fetal heart rate ranging from 120-160 bpm. Measurements was obtained from ≥ 4 consecutive flow velocity waveforms of good quality and averaged. From the flow velocity waveforms of the UA & MCA, the pulsatility index (PI) & the resistance index (RI) was measured. From the flow velocity waveforms of the DV, peak velocity index (PVIV), peak systolic velocity (PSV) and A wave was measured. From the umbilical vein flow, the presence or absence of pulsatile flow was recorded. All labours was attended by an expert neonatologist who was blinded to the results of Doppler indices measurements & the following was recorded: APGAR score at (1 & 5 min) - Neonatal birth weight (Fetal growth restriction will defined as birth weight of less than 10th percentile of newborn weight in normal pregnancies at corresponding gestational age) - the occurrence of respiratory complications [Transient Tachypnea of the newborn (TTN) or Respiratory Distress Syndrome (RDS)] - The further need for neonatal intensive care unit (NICU) admission & Perinatal death.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age (GA): 34 - 38weeks of gestations (confirmed by a reliable date for the last menstrual period or /and 1st trimester ultrasound scan).
* The current Pregnancy complicated with severe hypertension (gestational hypertension, preeclampsia, chronic hypertension and chronic hypertension with superimposed preeclampsia).
* Singleton living fetus.

Exclusion Criteria:

* Maternal medical disorders rather than hypertension.
* Fetal congenital anomalies.
* Rupture of membrane.
* Antepartum hemorrhage (placenta previa or accidental hemorrhage).
* The maternal administration of respiratory depressants within 2 hours from the delivery of the fetus (e. g., opioid analgesic )

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 60 pregnant women with singleton living fetus between 34 -38 wks gestation known to have severe hypertension in the current pregnancy were included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
The diagnostic value of umbilical artery (UA) Doppler indices (RI & PI) in predicting adverse perinatal outcome among severely hypertensive patients | within 24 hours before delivery and post natal
  sensitivity and specificity of umbilical artery RI & PI in detecting IUGR and APGAR score less than 7 at 5 minutes

SECONDARY OUTCOMES:
The diagnostic value of Middle cerebral artery (MCA) Doppler indices (RI & PI) in predicting adverse perinatal outcome among severely hypertensive patients | within 24 hours before delivery and post natal
  sensitivity and specificity of middle cerebral artery RI & PI in detecting IUGR and APGAR score less than 7 at 5 minutes
The diagnostic value of cerebro/placentaI Ratio in predicting adverse perinatal outcome among severely hypertensive patients. | within 24 hours before delivery and post natal
  sensitivity and specificity of of MCA/UA PI Ratio in detecting IUGR and APGAR score less than 7 at 5 minutes
The diagnostic value of Ductus Venousus Doppler indices in predicting adverse perinatal outcome among severely hypertensive patients. | within 24 hours before delivery and post natal
  sensitivity and specificity of peak velocity index (PVIV), peak systolic velocity (PSV) and abnormal A wave in detecting IUGR and APGAR score less than 7 at 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: moutaz elsherbini, MD, Principal Investigator — Assistant professor of obstetrics and gynecology
Locations (1):
- Kasr Elainy Hospital (Faculty of Medicine - Cairo University), Cairo, Egypt